CLINICAL TRIAL: NCT05687929
Title: Real-World Registry Study on Clinical Analgesic Effect of Acetylaconitine Tablets
Status: Recruiting | Type: Observational
Sponsor: Ke Ma (Other)
Responsible Party: Sponsor-Investigator, Ke Ma, Principal Investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: XH-22-008
Record Dates: First submitted 2022-12-27; First posted 2023-01-18 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To observe the clinical analgesic effect, safety and adverse reactions of acetylaconitine.
2. To study and analyze the main influencing factors of the acetylaconitine tablets.

DETAILED DESCRIPTION:
The outpatients/inpatients meeting the criteria are included into this study after signing the Informed Consent Form. The patients received 5 visits in total, which take place after the patients are included into the real-world study, on the 3rd day after enrollment and at the 1st, 4th, 8th and 12th weeks thereafter, in the form of outpatient follow-up, telephone follow-up and APP follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain > 1 month and VAS > 40 mm Patients who can take the acetylaconitine tablets orally

Exclusion Criteria:

* Patients who cannot communicate or receive follow-up Patients allergic to acetylaconitine Patients who have taken the acetylaconitine drugs orally

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic pain > 1 month and VAS > 40 mm Patients who can take the acetylaconitine tablets orally
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
VAS (0-100mm), IDpain | December 2022 to December 2023
  Pain score

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No